CLINICAL TRIAL: NCT05140447
Title: Temperature Change of the Pulpal Floor and Restoration With Preheated Resin Composite (A Randomized Clinical Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alshimaa Nasser Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Alshimaa Nasser Mahmoud, post grade student, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 490
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Preheating of Resin Composite
Keywords: preheating of resin composite; pulpal floor temperature; resin composite; BIS-GMA free resin composite; BIS-GMA containing resin composite; restoration temperature

STUDY DESIGN:
Intervention Model Description: Forty posterior teeth were randomly divided into two groups of 20 teeth. According to types of restorative materials used (A), the first group was restored by Bis-GMA free resin composite (A1) and the second group was restored by Bis-GMA containing resin composite (A2).
  Each group was subdivided into 2 subgroups of 10 teeth each according to preheating temperatures used (T), the first subgroup (T1) was preheated at 50◦ C and the second subgroup (T2) was preheated at 70◦ C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Admira 50º C (Active Comparator): in this subgroup the patient's teeth was restored with Admira fusion extra resin composite preheated to 50º C
  Interventions: Other: preheating of resin composite
- Admira 70º C (Active Comparator): in this subgroup the patient's teeth was restored with Admira fusion extra resin composite preheated to 70º C
  Interventions: Other: preheating of resin composite
- Viscalor 50º C (Active Comparator): in this subgroup the patient's teeth was restored with Viscalor resin composite preheated to 50º C
  Interventions: Other: preheating of resin composite
- Viscalor 70º C (Active Comparator): in this subgroup the patient's teeth was restored with Viscalor resin composite preheated to 70º C
  Interventions: Other: preheating of resin composite

INTERVENTIONS:
Other: preheating of resin composite — evaluate the effect of preheating BIS-GMA free resin composite at different temperatures on temperature change of the pulpal floor and restorations and compare it with BIS-GMA containing resin composite.
  Other Names: warming of resin composite

SUMMARY:
clinical evaluation of the effect of preheating BIS-GMA free resin composite at different temperatures on temperature change of the pulpal floor and restorations and compare it with BIS-GMA containing resin composite.

Hypothesis: Could the preheated composite affect the temperature of the pulpal floor

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women patients of 25-45 years.
* They should have a good oral hygiene level.
* Presence of at least two posterior class I or II carious lesions to be restored with two different composite resin restorations.
* All carious lesions in selected patients didn't close to the pulp in the preoperative radiograph.
* No preoperative pain.
* Normal occlusal contact with opposing teeth.
* No history of periodontal treatment, including periodontal surgery, in the past year.
* All patients had to sign a written consent before being included.
* A good likelihood of recall availability.

Exclusion Criteria:

* patient with severe periodontitis or severe erosion damage.
* patients with a compromised medical history or had received therapeutic irradiation to the head and neck region.
* If analgesics or antibiotics had administered by the patient during the past 12 hours preoperatively as it might alter their pain perception.
* patients reported bruxism or clenching.
* Greater than grade I mobility or pocket depth greater than 5mm.
* Non-restorable teeth or hopeless teeth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption.
* Alcoholic and smoker patients.
* Pregnant or breastfeeding ladies.
* Patients who had physical disabilities, or who are unable to brush their teeth.
* Individuals who had sensitive teeth but with one of the following conditions was excluded from the study, teeth with large restoration, abutment of teeth of removable partial dentures, dental restorations, abutment of teeth of removable partial dentures, enamel cracks, leakage of fillings or other restorations teeth, dental pulp lesions, dental abscesses, pulpitis, and atypical facial pain.
* Patients who had non-carious lesions like attrition, erosion, abrasion or abfraction.
* Patients had participated in a clinical trial within 6 months before commencement of this trial.
* Patients unable to return for a recall appointment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
pulpal floor temperature and restoration temperature | one year
  evaluation the effect of preheating BIS GMA free resin composite at different temperature on temperature change of pulpal floor and restoration and compare it with BIS GMA containing resin composite
  All readings were taken with the presence of a rubber dam and recorded in Celsius (°C).
  Five temperature readings were measured for each tooth; (C0): pulpal floor temperature before beginning the restorative procedure. (C1): pulpal floor temperature during placement of preheated composite. (C2): top composite surface after packing and before curing. (C3): pulpal floor temperature after curing of the preheated composite. (C4): top composite surface after curing. The pulpal floor and the restoration temperature of each tooth was measured by a K-type temperature Probe attached to portable mini type thermometer device

SECONDARY OUTCOMES:
The effect of different preheating temperatures on restoration temperature and pulpal floor temperature | one year
  Five temperature readings were measured for each tooth; (C0): pulpal floor temperature before beginning the restorative procedure. (C1): pulpal floor temperature during placement of preheated composite. (C2): top composite surface after packing and before curing. (C3): pulpal floor temperature after curing of the preheated composite. (C4): top composite surface after curing. The pulpal floor and the restoration temperature of each tooth was measured by a K-type temperature Probe attached to portable mini type thermometer device

OTHER OUTCOMES:
The difference in restoration and pulpal floor temperatures before and after curing of preheated resin composite | one year
  Five temperature readings were measured for each tooth; (C0): pulpal floor temperature before beginning the restorative procedure. (C1): pulpal floor temperature during placement of preheated composite. (C2): top composite surface after packing and before curing. (C3): pulpal floor temperature after curing of the preheated composite. (C4): top composite surface after curing. The pulpal floor and the restoration temperature of each tooth was measured by a K-type temperature Probe attached to portable mini type thermometer device

CONTACTS AND LOCATIONS:
Overall Officials: Mona I Riad, Professor, Study Director — Professor at Faculty of Dentistry Cairo University; Nermin A Mahmoud, Lecturer, Study Director — Lecturer at Faculty of Dentistry Minia University
Locations (1):
- Faculty of Dentistry - Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes